CLINICAL TRIAL: NCT07379879
Title: Acute Neurochemical and Cognitive Responses to High Intensity Interval Training vs. Moderate- and Low-Intensity Continuous Training in Young Adult Males
Brief Title: Acute Neurochemical and Cognitive Changes After HIIT vs MICT/LICT
Acronym: ANCCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, serkan pancar, Assoc. Prof., Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 185-8/10
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: BDNF; Cognitive Performance; Lactate; Exercise Intensity
Keywords: BDNF; Cognitive Performance; Stroop Test
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants remained seated quietly at rest for 24 minutes in a quiet, well-lit room, matched to the exercise sessions for time schedule and environmental conditions. No physical activity was performed during this period.
- Low-intensity continuous training (Experimental): They were asked to perform low intensity exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: Low Intensity Exercise
- Moderate-intensity continuous training (Experimental): They were asked to perform moderate intensity exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: Moderate-Intensity Continuous Exercise
- High-intensity interval training (Experimental): They were asked to perform HIIT exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Behavioral: Low Intensity Exercise — Participants ran continuously for 24 minutes at 50-60% of their MAS without rest
  Arms: Low-intensity continuous training
Behavioral: Moderate-Intensity Continuous Exercise — Participants completed a continuous 24-min running bout at 70-80% of their MAS. The exercise was performed at a steady, uninterrupted pace throughout the session, with no planned rest periods. Participants were instructed to maintain the prescribed pace for the entire duration
  Arms: Moderate-intensity continuous training
Behavioral: High-Intensity Interval Training — Participants performed 15-s running bouts at 110-120% of MAS, with the target distance for each bout pre-calculated from individual MAS (speed × time). Running was conducted shuttle-style between two cones. At the whistle, participants ran from one cone to the other for 15 s and then remained standing still for a 15-s passive rest at that cone. At the next whistle, they ran back in the opposite direction, followed by another 15-s stationary recovery. This 15-s run/15-s recovery cycle continued for 3 min, constituting one set (6 runs and 6 recovery intervals per set). Four sets were completed, separated by 3-min passive inter-set rest, resulting in a total session duration of 24 min
  Arms: High-intensity interval training

SUMMARY:
This study examines whether the intensity of a single running session changes a blood marker related to brain health (brain-derived neurotrophic factor, BDNF), blood lactate, and performance on a short thinking task that measures attention and self-control (the Stroop test) in healthy young adult men.

Twelve healthy males (18-25 years) will complete four separate sessions in a randomized, counterbalanced order, with at least 7 days between sessions. Each session includes an 8-minute warm-up followed by 24 minutes of one of the following conditions: low-intensity continuous running, moderate-intensity continuous running, high-intensity interval running (repeated 15-second fast runs with 15-second passive rest, organized into sets), or a seated rest control session. Running pace will be individualized based on a prior fitness test.

A small venous blood sample (about 8 mL) will be collected immediately before and within 1 minute after each session. After each session, participants will complete the Stroop test. The main outcomes are the before-to-after changes in serum BDNF, blood lactate, and Stroop test performance across the four conditions.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 25 years
* No known medical condition that prevents participation in exercise
* Not currently using any pharmacological agents

Exclusion Criteria:

* Experiencing any discomfort before, during, or after exercise
* Current or past diagnosis of pharmacological or doping substance use
* Engaging in regular exercise (more than 3 times per week) within the last 2 weeks
* History of alcohol or substance addiction
* Any other condition or factor that may prevent full participation in the study protocol

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants were eligible to participate in this study based on biological sex.
Enrollment: 12 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Lactate | Baseline, Immediately After Exercise (Day 1)
  Lactate levels were measured in millimoles per liter (mmol/L) from capillary/venous blood samples taken before and after exercise using a lactate analyzer.
BDNF | Baseline, Immediately After Exercise (Day 1)
  BDNF levels were measured using a Sunred brand ELISA kit from blood samples taken baseline and after exercise, and the results were reported in ng/mL units.
Stroop Test | Baseline and immediately after exercise (Day 1)
  Stroop test performance will be assessed as an indicator of executive function, primarily selective attention and inhibitory control. In this task, participants are required to identify the ink color of presented stimuli while suppressing the automatic tendency to read the written word, particularly during incongruent trials (e.g., the word "red" printed in blue ink). The test will be administered immediately after each session. Outcomes will include reaction time and accuracy (and/or an interference score derived from incongruent vs. congruent conditions). Reaction time will be recorded in seconds (s), with poorer performance reflected by slower responses and/or more errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A key risk is participant re-identification due to the small sample size and the presence of biomarker and performance data that could enable triangulation, even after de-identification.